CLINICAL TRIAL: NCT05583253
Title: Visual Outcome of Small Gauge Pars-plana Vitrectomy for Retinal Detachment With Previous Refractive Surgery
Brief Title: Visual Outcome of Vitrectomy After Refractive Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Assistant professor of Ophthalmology, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rc 12-2022
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Retinal Detachment; Refractive Errors
MeSH Terms: conditions — Retinal Detachment; Refractive Errors | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitrectomy group with previous refractive surgery (Active Comparator): Cases with primary retinal detachment that are prepared for pars-plana vitrectomy with previous history of refractive surgery.
  Interventions: Procedure: Vitrectomy
- Vitrectomy group with no previous intraocular surgery (Active Comparator): Subjects with primary retinal detachment that are prepared for pars-plana vitrectomy with no previous history of intraocular surgery.
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy — Small gauge pars-plana vitrectomy for management of retinal detachment.
  Other Names: Pars-plana vitrectomy

SUMMARY:
Results of retinal detachment surgery may be affected in cases with history of previous intraocular surgery.

DETAILED DESCRIPTION:
Pars-plana vitrectomy for management of retinal detachment has favorable visual outcome with early intervention and development of small gauge instruments, cases with previous refractive surgery may be affected by other factors that may change the final visual outcome.

In this study, we aim to analyze the effect of refractive surgeries on the final visual outcome after vitrectomy for the management of retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* cases diagnosed with primary retinal detachment and prepared for pars-plana vitrectomy.
* cases with previous history for refractive surgery were enrolled in refractive surgery group.

Exclusion Criteria:

* cases with corneal diseases or trauma that may affect the final visual outcome.
* cases with other retinal diseases that may affect the final visual outcome as age related macular degenerations and diabetic eye disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Baseline and 6 months after surgery.
  Changes in visual acuity from baseline and at the 6th month of follow-up measured by snellen chart and converted to logMAR units for statistical analysis.

SECONDARY OUTCOMES:
Corneal endothelial cells count | Baseline and 6 months after surgery.
  Changes in corneal endothelial cells counts measured by specular microscopy in cells/millimeters2 units.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa A Abdelshafy, MD, Study Director — Benha University
Locations (1):
- Benha University, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: No